CLINICAL TRIAL: NCT00388960
Title: Randomized Phase II Study of Amrubicin as Single Agent or in Combination With Cisplatin Versus Etoposide-cisplatin as First-line Treatment in Patients With Extensive Stage SCLC (ES)
Brief Title: Study of Amrubicin With or Without Cisplatin Versus Etoposide-cisplatin for Extensive Stage Small Cell Lung Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Celgene (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: EORTC Protocol 08062; 2006-001956-11 (EudraCT Number); NCT00424073 (obsolete NCT alias)
Record Dates: First submitted 2006-10-13; First posted 2006-10-17 (Estimated); Last update posted 2019-11-19 (Actual); Status verified 2019-11

CONDITIONS: Small Cell Lung Cancer
Keywords: small cell lung cancer; amrubicin
MeSH Terms: conditions — Small Cell Lung Carcinoma | interventions — amrubicin; Cisplatin; Etoposide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Amrubicin (Experimental): Amrubicin 45mg/m<2> IV days 1, 2, 3 of each 21-day cycle until disease progression.
  Interventions: Drug: Amrubicin
- Amrubicin plus Cisplatin (Experimental): Amrubicin 40mg/m<2> IV days 1, 2, 3 plus cisplatin 60mg/m<2> IV day 1 of each 21-day cycle until disease progression.
  Interventions: Drug: Amrubicin; Drug: Cisplatin
- Cisplatin plus etoposide (Active Comparator): Cisplatin 75mg/m<2> IV day 1 plus etoposide 100mg/m<2> IV day 1 and 200mg/m<2> orally days 2, 3 or etoposide 100mg/m<2> IV days 1, 2, 3 each 21-day cycle until disease progression.
  Interventions: Drug: Cisplatin; Drug: Etoposide

INTERVENTIONS:
Drug: Amrubicin — Amrubicin 45mg/m<2> IV days 1, 2 3 of each 21-day cycle until disease progression.
  Amrubicin 40mg/m<2> IV days 1, 2, 3 plus cisplatin 60mg/m<2> day 1 of each 21-day cycle until disease progression.
  Arms: Amrubicin; Amrubicin plus Cisplatin
Drug: Cisplatin — Amrubicin 40mg/m<2> IV days 1, 2, 3 plus Cisplatin 60mg/m<2> day 1 of each 21-day cycle until disease progression.
  Cisplatin 75mg/m<2> IV day 1 plus etoposide 100mg/m<2> IV day 1 and 200mg/m<2> orally days 2, 3 or etoposide 100mg/m<2> IV days 1, 2, 3 of each 21-day cycle until disease progression.
  Arms: Amrubicin plus Cisplatin; Cisplatin plus etoposide
Drug: Etoposide — Cisplatin 75mg/m<2> IV day 1 plus etoposide 100mg/m<2> IV day 1 and 200mg/m<2> orally days 2, 3 or etoposide 100mg/m<2> IV days 1, 2, 3 of each 21-day cycle until disease progression.
  Arms: Cisplatin plus etoposide

SUMMARY:
The purpose of the study is to document the activity and safety of single agent amrubicin, amrubicin combined with cisplatin, and etoposide combined with cisplatin as first-line treatment in extensive disease small cell lung cancer.

ELIGIBILITY:
Inclusion Criteria:

* Histologically/cytologically proven small cell lung cancer
* Extensive disease
* Measurable disease
* World Health Organization (WHO) performance status 0-2
* Age 18 years or older
* Normal baseline cardiac function
* No prior systemic chemotherapy for small cell lung cancer
* Adequate organ function including bone marrow, kidney, and liver
* No history of interstitial lung disease or pulmonary fibrosis
* No history of prior malignancy unless patient has been disease free for greater than 5 years, or the tumour was a non-melanoma skin cancer or in-situ carcinoma of the cervix
* No pregnancy or breast feeding; patients of child-bearing potential must agree to use an appropriate method of contraception
* Written informed consent before randomization

Exclusion criteria:

* Pre-existing peripheral neuropathy (greater than Grade 1, CTCAE version 3.0)
* Uncontrolled or severe cardiovascular disease
* Any psychological, familial, sociological or geographical condition potentially hampering compliance with the study protocol and follow-up schedule

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 99 (Actual)
Dates: Start 2006-11-01 (Actual); Primary Completion 2010-04-01 (Actual); Study Completion 2010-12-01 (Actual)

PRIMARY OUTCOMES:
Objective tumor response rate according to RECIST criteria measured every 2 cycles (every 6 weeks) | Until Disease Progression

SECONDARY OUTCOMES:
Toxicity | Until 30 days after last protocol treatment
Progression-free survival | Until disease progression or death
Overall survival | Until death

CONTACTS AND LOCATIONS:
Overall Officials: Mary O'Brien, MD, Principal Investigator — Royal Marsden Hospital, London, UK
Locations (25):
- Belgium (7):
  - Algemeen Ziekenhuis Middelheim, Antwerp
  - Universitair Ziekenhuis Antwerpen, Edegem
  - Universiteit Gent, Ghent
  - U.Z. Gasthuisberg, Leuven
  - Domaine Universitaire du Sart-Tilman, Liège
  - Centre Hospitalier Regional de la Citadelle, Liège
  - Clinique Sainte Elisabeth, Namur
- Italy (2):
  - Instituto Nazionale per la Ricerca sul Cancro, Genova
  - Universita Degli Studi Di Udine, Udine
- Netherlands (6):
  - Academisch Medisch Centrum, Amsterdam
  - The Netherlands Cancer Institute Antoni Van Leeuwenhoekziekenhuis, Amsterdam
  - Medisch Spectrum Twente - Dept of Pulmonary Diseases, Enschede
  - Leiden University Medical Centre, Leiden
  - Academisch Ziekenhuis Maastricht, Maastricht
  - Isala Kliniek, Zwolle
- Medical University of Gdansk - Dept Radiotherapy, Gdansk, Poland
- United Kingdom (9):
  - Clatterbridge Centre for Oncology NHS Trust, Bebington, Merseyside
  - University of Dundee - Ninewells Hospital, Dundee, Scotland
  - Belfast City Hospital, Belfast
  - Western General Hospital, Edinburgh
  - Princess Royal Hospital, Hull
  - Royal Marsden Hospital, London, London
  - Christie Hospital, Manchester
  - Sir Bobby Robson Cancer Trials Research Centre, Newcastle upon Tyne
  - Royal Marsden Hospital Lung Unit, Sutton

REFERENCES:
- [Background] O'Brien ME, Konopa K, Lorigan P, Bosquee L, Marshall E, Bustin F, Margerit S, Fink C, Stigt JA, Dingemans AM, Hasan B, Van Meerbeeck J, Baas P. Randomised phase II study of amrubicin as single agent or in combination with cisplatin versus cisplatin etoposide as first-line treatment in patients with extensive stage small cell lung cancer - EORTC 08062. Eur J Cancer. 2011 Oct;47(15):2322-30. doi: 10.1016/j.ejca.2011.05.020. Epub 2011 Jun 16. PMID 21684151
- [Background] Liddell RP, Evans NS. May-Thurner syndrome. Vasc Med. 2018 Oct;23(5):493-496. doi: 10.1177/1358863X18794276. No abstract available. PMID 30187833